CLINICAL TRIAL: NCT06982183
Title: The Effects of Propranolol, Hydrocortisone, and Morphine on Military-Relevant Performance Outcomes: A Randomized, Blinded, Placebo Controlled Study
Brief Title: The Effects of Propranolol, Hydrocortisone, and Morphine on Military-Relevant Performance Outcomes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WRAIR #2950; MO210072 (Other Grant/Funding Number: USAMRDC Military Operational Medicine Research Program (MOMRP))
Record Dates: First submitted 2025-05-01; First posted 2025-05-21 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Fear of Spiders; Acute Stress Reaction
Keywords: Fear of Spiders; morphine; propranolol; hydrocortisone; randomized controlled trial; neuropsychological tests; acute stress reaction
MeSH Terms: conditions — Arachnophobia; Stress Disorders, Traumatic, Acute | interventions — Propranolol; Hydrocortisone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Propranolol (oral) (Active Comparator)
  Interventions: Drug: Propranolol
- Placebo (oral) (Placebo Comparator)
  Interventions: Drug: Placebo (oral)
- Hydrocortisone (IM) (Active Comparator)
  Interventions: Drug: Hydrocortisone
- Morphine (IM) (Active Comparator)
  Interventions: Drug: Morphine
- Placebo (IM) (Placebo Comparator)
  Interventions: Drug: Placebo (IM)

INTERVENTIONS:
Drug: Propranolol — An administration of a 40-mg propranolol capsule immediately after tarantula exposure
  Arms: Propranolol (oral)
Drug: Hydrocortisone — An intramuscular administration of 62.5 mg/1 ml of hydrocortisone immediately after tarantula exposure
  Arms: Hydrocortisone (IM)
Drug: Morphine — An intramuscular administration of 5 mg/1 ml of morphine immediately after tarantula exposure
  Arms: Morphine (IM)
Drug: Placebo (oral) — An administration of a placebo capsule after tarantula exposure
  Arms: Placebo (oral)
Drug: Placebo (IM) — An intramuscular administration of 1 ml of saline immediately after tarantula exposure
  Arms: Placebo (IM)

SUMMARY:
This clinical trial aims to evaluate the nature and duration of effects of three FDA-approved medications (propranolol, hydrocortisone, and morphine) on military-relevant cognitive, emotional, and motor performance following an exposure to a stressful situation (i.e., exposure to a tarantula) in physically healthy adult volunteers (aged 18 - 40) with fear of spiders to help the future development of medications for treating Acute Stress Reactions.

The main questions this study aims to answer are:

Will placebo treatment (oral placebo) result in significant decrements in Psychomotor Vigilance Task (PVT) performance compared to propranolol treatment?

Will placebo treatment [intramuscular (IM) placebo] result in significant decrements in PVT performance compared to hydrocortisone treatment?

Will placebo treatment (IM placebo) result in significant decrements in PVT performance compared to morphine treatment?

Participants will receive one of five study medications (oral propranolol, oral placebo, IM hydrocortisone, IM morphine, or IM morphine) after a brief exposure to a tarantula. Participants will complete cognitive and simple motor tasks and psychological assessments before and after the study medication administration.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-lactating females 18 to 40 (inclusive) years of age.
* Females of child-bearing potential must be on some form of birth control, if sexually active (e.g., oral contraceptive, condom, intrauterine device, etc.)
* Score of 80% or greater on a "Volunteer Comprehension Assessment" test.
* Score equal to or greater than 54 on the Fear of Spiders Questionnaire.
* Body weight between 91 and 250 pounds (inclusive).
* Live close enough to be able to commute to Walter Reed Army Institute of Research during the study participation.

Exclusion Criteria:

* Contraindications due to study medications, including a history of allergic/hypersensitivity reactions to a beta blocker, an opiate agonist or a steroid, or a history of other adverse reactions to these classes of drugs (such as an episode of steroid psychosis).
* A history of allergic reactions to a spider bite.
* A history of abuse or addiction to illicit drugs (including marijuana) or prescribed medication (e.g., opioid) (diagnosed or suspected based on the medical history).
* Use a nicotine product (e.g., cigarette, cigar, vape) more than 3 days per week.
* Self-reported caffeine use in excess of 600 mg (e.g., approximately 10 caffeinated sodas or approximately 29 ounces of brewed coffee) per day on average or not being able to go without caffeine during the In-Lab visits.
* History of neurologic disorder (to include but not limited to epilepsy, hydrocephalus, MS). An infrequent or resolved single neurological event (e.g., childhood seizure, rare sporadic migraine headaches, resolved meningeal infection with no sequelae) or a history of mild traumatic brain injury may be deemed non-exclusionary at the discretion of the examining study medical investigator
* Score of 10 or above on the Beck Depression Inventory (BDI) or a score of > 0 on item 9 "Suicidal Thoughts or Wishes" of the BDI
* Score of 41 or above on the State-Trait Anxiety Inventory - Trait (STAI-T).
* Score of 20 or above on the PROMIS Emotional Distress - Anxiety - Short Form.
* Score of 33 or above on the PTSD Checklist, 5th Edition (PCL-5)
* History of cardiovascular disease (to include but not limited to arrhythmias, valvular heart disease, congestive heart failure, history of sudden cardiac death or myocardial infarction).
* A history of asthma or any type of reactive airways disease or any acute or chronic pulmonary disorder that could lead to a compromise of blood oxygenation in the setting of a modest reduction in tidal volume or respiratory rate, to include neuromuscular disorders.
* Regularly work night shifts or have a habitual sleep/wake schedule that is not conducive to compliance with the recommended sleep time (11:00 pm - 6:00 am) during participation (e.g., extremely early or late habitual bedtime or rise time, to be determined on a case-by-case basis by the principal investigator or an associate investigator).
* A diagnosis of sleep apnea.
* Kidney disease or kidney abnormalities, liver disease or liver abnormalities, or any other metabolic derangements (endocrine disorders, hyperglycemia, etc.) that could alter neurophysiological function.
* Liver disease or significant liver abnormalities as determined by examining study medical investigator.
* Self-reported history of hospitalization for a psychiatric disorder within the past year or with a previous history of a psychotic, bipolar disorder or personality disorder. For a history of a diagnosis of any other psychiatric disorder, a potential participant's symptoms must either be resolved to a degree that a diagnosis is no longer applied or their symptoms must have been stabilized by pharmacological or nonpharmacological treatments for a period of at least 90 days or greater as deemed exclusionary or non-exclusionary at the discretion of the examining study medical investigator.
* Self-reported or suspected current use of antipsychotics, anticonvulsants, or mood stabilizers, to be determined on a case-by-case basis by the examining study medical investigator.
* Self-reported or suspected current use of products or drugs that have CNS depressant effects, to be determined on a case-by-case basis by the examining study medical investigator.
* Self-reported or suspected use of products or drugs that cannot be safely discontinued during in-laboratory phases, to be determined on a case-by-case basis by the examining study medical investigator.
* Self-reported or suspected current heavy alcohol use (minimum limit to define heavy alcohol use is 14 drinks per week for males and 7 drinks per week for females or as determined by the examining study medical investigator).
* (Females only) Positive urine pregnancy result
* (Females only) Self-reported or suspected current breast-feeding or collecting breast-milk.
* Resting blood pressure above 140/90 or resting pulse > 110 beats per minute. Note that if a repeat measurement is within range, the volunteer will not be excluded.
* Resting blood pressure below 100/60 or pulse oxygenation <92%. Volunteers with a resting pulse < 60 bpm will be excluded unless a history of regular vigorous aerobic exercise and findings on the physical examination (including BMI) suggest a high level of cardiovascular fitness, in which case a resting pulse in the range of 50 - 59 bpm may not be exclusionary.
* BMI ≥ 31. The inclusion of individuals with BMI between 30 and 31 (Obese Class I) will be determined using medical investigator's discretion.
* Clinically significant values (as determined by the reviewing study medical investigator) for any hematology or chemistry parameter. Reviewing study medical investigator may opt to repeat any clinically significant tests and include volunteers whose repeat test values are not clinically significant.
* Currently on or recently ended immunotherapy (e.g., allergy shots).
* Have taken a vaccine within 30 days prior to enrollment to the study. For volunteers who report recently taking a vaccine during the screening visit, their In-Lab Day 1 visit will be scheduled at least 30 days after the date of the most recent vaccination.
* Positive urine drug result during screening visit or In-Lab Days 1- 2; Exhibiting behaviors consistent with illicit drug use on In-Lab Day 3.
* Positive saliva alcohol result during screening visit or In-Lab Days 1-3.
* Inability to read and sign consent.
* Failure to obtain required approved official leave to participate (federal civilian employees and active duty military only)
* Failure to cooperate with requirements of the study
* Failure to provide viable emergency contact(s) for the duration of the study
* Self-reported or suspected current use of illicit drugs (including but not limited to benzodiazepines, amphetamines, cocaine, marijuana).
* Current use and/or prescription for opioid, steroid or anti-hypertensive and/or any medication the Medical Investigator deems would interact adversely with study compounds.
* Current use of medications that can adversely interact with propranolol, hydrocortisone and/or morphine to include anti-depressants that are cytochrome P450 2D6 inhibitors.
* Current diabetes.
* GI disorders - motility disorders
* Failure to pass certain tests
* Failure to provide a social security number or tax identification number in order to be paid for screening and participation in the study.
* Current participation in another ongoing clinical trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Psychomotor Vigilance Task | Baseline and post-treatment time points within approximately 25 hours following the study medication administration.
  Measure of cognitive performance. Reaction time (millisecond)

SECONDARY OUTCOMES:
Behavioral Approach Task | Baseline and approximately 24 hours post-treatment.
  An behavioral assessment to examine how closely individuals can approach an aversive stimulus.
Go/No-Go task | Baseline and post-treatment time points within approximately 25 hours following the study medication administration.
  Measure of cognitive performance.
Matching to Sample task | Baseline and post-treatment time points within approximately 25 hours following the study medication administration.
  Measure of cognitive performance
Simple Reaction Time task | Baseline and post-treatment time points within approximately 25 hours following the study medication administration.
  Measure of cognitive performance.
The Automated Neuropsychological Assessment Metrics (ANAM) Mood Scale | Baseline and post-treatment time points within approximately 25 hours following the study medication administration.
  Measure of mood.
WRAIR Mood Battery | Baseline and post-treatment time points within approximately 25 hours following the study medication administration.
  A short battery of measures of various aspects of mood.
Heart rate | Before, during, and after behavioral approach task and aversive stimulus exposure. 30 minutes - 1 hour at each time point.
  Continuous measure of heart rate.
Biosway | Baseline and post-treatment time points within approximately 25 hours following the study medication administration.
  Measure of motor performance
Triple Hop Test | Baseline and post-treatment time points within approximately 25 hours following the study medication administration.
  Measure of motor performance.
Drug Effects Questionnaire | Multiple time points within approximately 25 hours following the study medication administration.
  Measure of subjective response to a substance.
Subjective Fear Scale | Baseline, during the behavioral approach test and aversive stimulus exposure, and time points within approximately 25 hours after the study medication administration.
  Subjective measure of fear. A 0 - 100 numerical scale.
Subjective Anxiety Scale | Baseline, during the behavioral approach test and aversive stimulus exposure, and time points within approximately 25 hours after the study medication administration.
  Subjective measure of anxiety. A 0 - 100 numerical scale.
Subjective Stress Scale | Baseline, during the behavioral approach test and aversive stimulus exposure, and time points within approximately 25 hours after the study medication administration.
  Subjective measure of stress. A 0 - 100 numerical scale.
Symptom checklist | Baseline, pre-medication administration, and time points within approximately 27 hours after the medication administration.
  Checklist to capture adverse drug reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Research Center (SRC), Walter Reed Army Institute of Research, Silver Spring, Maryland, United States